CLINICAL TRIAL: NCT00545909
Title: A Randomised, Open Label Study to Investigate the Impact of Bone Marker Feedback at 2 Months on Adherence to Monthly Oral Bonviva (Ibandronate) in Women With Post-menopausal Osteoporosis.
Brief Title: BEATRIS Study: A Study of Adherence to Bonviva (Ibandronate) Once Monthly in Women With Post-Menopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19913
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Active Comparator)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 6 months (+ feedback)
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 6 months (- feedback)
  Arms: 2

SUMMARY:
This 2 arm study will assess the impact of Bone Marker Feedback (BMF), using blood sampling and communication of the results at 2 months, on adherence to monthly Bonviva (150mg po) in women with post-menopausal osteoporosis. Patients will be randomized into either 1) a group which receives bone marker feedback or 2)a group which does not receive feedback on the results. The study will also assess patient satisfaction with treatment with once monthly Bonviva. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory post-menopausal women with osteoporosis;
* 55-85 years of age;
* eligible for bisphosphonate treatment;
* naive to bisphosphonate therapy, or lapsed users (last bisphosphonate intake > 6 months ago).

Exclusion Criteria:

* inability to stand or sit in an upright position for at least 60 minutes;
* inability to swallow a tablet whole;
* hypersensitivity to bisphosphonates;
* administration of any drug, or presence of active disease, known to influence bone metabolism;
* uncorrected hypocalcemia or other bone disturbances of bone and mineral metabolism;
* history of major upper gastrointestinal disease.

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Comparison of percentage of patients with >=83% adherence to Bonviva in feedback vs no feedback group | 6 months

SECONDARY OUTCOMES:
Patient satisfaction by OPSAT-Q and OPPS. | 6 months
Tolerability; SAEs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- Austria (7):
  - Bregenz
  - Graz
  - Innsbruck
  - Linz
  - Salzburg
  - Vienna
  - Vöcklabruck
- Belgium (28):
  - Aalst
  - Antwerp
  - Aye
  - Braine-l'Alleud
  - Bruges
  - Brussels
  - Charleroi
  - Dinant
  - Ekeren
  - Genk
  - Ghent
  - Godinne
  - Hasselt
  - Jambes
  - Knokke
  - Kortrijk
  - La Louvière
  - Liège
  - Mechelen
  - Merksem
  - Mons
  - Ostend
  - Roeselare
  - Sijsele
  - Tournai
  - Turnhout
  - Waremme
  - Wilrijk
- Greece (4):
  - Athens
  - Kifissia
  - Larissa
  - Thessaloniki
- Ireland (2):
  - Gorey
  - Tipperary
- Luxembourg, Luxembourg